CLINICAL TRIAL: NCT01491815
Title: A Multicenter, Randomized, Open-label, Blinded-assessor, Phase 4 Study in Patients With Early Rheumatoid Arthritis to Compare Active Conventional Therapy Versus Three Biologic Treatments, and Two De-escalation Strategies in Patients Who Respond to Treatment
Brief Title: Active Conventional Therapy Compared to Three Different Biologic Treatments in Early Rheumatoid Arthritis With Subsequent Dose Reduction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ronald van Vollenhoven, prof., Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NORD-STAR; 2011-004720-35 (EudraCT Number); 2011/2069-31/4 (Other: Regional Ethical Review Board)
Record Dates: First submitted 2011-12-08; First posted 2011-12-14 (Estimated); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol; Abatacept; tocilizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Active conventional therapy (ACT) (Active Comparator): Non-biological DMARD's: Methotrexate plus steroids or Methotrexate plus Sulphasalazine and Hydroxychloroquine and steroids
  Interventions: Drug: Non-biological DMARD's
- Biologic agent 1 (Active Comparator): Cimzia: Certolizumab-pegol plus Methotrexate and steroids
  Interventions: Biological: Cimzia
- Biologic agent 2 (Active Comparator): Orencia: Abatacept plus Methotrexate and steroids
  Interventions: Biological: Orencia
- Biologic agent 3 (Active Comparator): RoActemra: Tocilizumab plus Methotrexate and steroids
  Interventions: Biological: RoActemra

INTERVENTIONS:
Drug: Non-biological DMARD's — Methotrexate: 25mg/week. SSZ: 2 g/day. HCQ: 35 mg/kg/week (Finland and Denmark) Methotrexate: 25mg/week. Prednisolone 20 mg/day tapered in 9 weeks to 5 mg/day, discontinued after 9 months. (Sweden, Norway, Iceland, and the Netherlands)
  Arms: Active conventional therapy (ACT)
Biological: Cimzia — Certolizumab-pegol: 200 mg s.c. every other week. Methotrexate: 25mg/week
  Arms: Biologic agent 1
Biological: Orencia — Abatacept: 125 mg s.c. every week. Methotrexate: 25mg/week
  Arms: Biologic agent 2
Biological: RoActemra — Tocilizumab is given as 4-weekly infusions at dosage 8 mg/kg or 162 mg in solution s.c. every week.
  Methotrexate: 25mg/week
  Arms: Biologic agent 3

SUMMARY:
This is an international (Sweden, Finland, Norway, Denmark, Iceland and the Netherlands) trial designed to compare the safety and efficacy of active conventional therapy (ACT) and three biologic treatments in subjects with early rheumatoid arthritis (RA). The global aim of this study is to assess and compare

1. the proportion of subjects who achieve remission with ACT versus three different biologic therapies (Certolizumab-pegol, Abatacept or Tocilizumab)
2. two alternative de-escalation strategies in patients who respond to first-line therapy.

DETAILED DESCRIPTION:
After completed enrollment a total of 812 patients were included in the study.

371 of the included patients have entered treatment part 2, 256 patients have exited the study after treatment part 1, 207 patients have had early termination and 322 patients have completed the full study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years of age.
2. Subject has a diagnosis of RA as defined by the newly established ACR/EULAR criteria, 2010. (Patients should also be classified according to the 1987-revised ACR-classification criteria, without this being an inclusion criteria).
3. <24 months from arthritis symptom debut (symptom duration will be registered).
4. Subject must have DAS28 (CRP) > 3.2.
5. ≥ 2 swollen joints AND ≥ 2 tender joints.
6. Subject must fulfill one of the following three criteria: RF positive OR ACPA positive OR CRP >10 mg/L.
7. Female subject is either not of childbearing potential (postmenopausal, surgically sterile etc.), or is of childbearing potential and practicing one of the following methods of birth control throughout the study and for 150 days after study completion:

   * Intrauterine device (IUD)
   * Contraceptives (oral, parenteral, patch) for three months prior to study drug administration)
   * A vasectomized partner
8. Female subjects of childbearing potential must have a negative serum pregnancy test at the Screening visit.
9. Subject is judged to be in good general health as determined by the principal investigator based upon the results of medical history, laboratory profile, physical examination, chest X-ray (CXR), and 12-lead electrocardiogram (ECG) performed at Screening.
10. Subjects must be able and willing to provide written informed consent and comply with the requirements of this study protocol.
11. Subjects must be able and willing to self-administer s.c. injections or have a qualified person available to administer s.c. injections.

Exclusion Criteria:

1. Subject has been previously treated with disease modifying antirheumatic drugs (DMARDs) for rheumatic diseases.
2. Current active inflammatory joint disease other than RA.
3. Subjects has had a dose of prednisone (or equivalent) >7.5 mg/day or has had a dose change within the preceding 4 weeks.
4. Subject has been treated with intra-articular or parenteral administration of corticosteroids in the preceding 4 weeks. Inhaled corticosteroids for stable medical conditions are allowed.
5. Subject has undergone joint surgery within the preceding two months (at joints to be assessed within the study).
6. Subject has chronic arthritis diagnosed before age 17 years.
7. Subject has a history of an allergic reaction or significant sensitivity to constituents of study drugs.
8. Subject has been treated with any investigational drug within one month prior to screening visit.
9. Active infection of any kind (excluding fungal infections of nail beds), or any major episode of infection requiring hospitalization within 4 weeks of screening.
10. Subject has a poorly controlled medical condition, such as uncontrolled diabetes, unstable heart disease, congestive heart failure, recent cerebrovascular accidents and any other condition which, in the opinion of the investigator, would put the subject at risk by participation in the study.
11. Subject has a history of clinically significant hematologic (e.g., severe anemia, leukopenia, thrombocytopenia), renal or liver disease (e.g., fibrosis, cirrhosis, hepatitis).
12. Subject has history of neurologic symptoms suggestive of central nervous system (CNS) demyelinating disease and/or diagnosis of central demyelinating disease.
13. Subject has history of cancer or lymphoproliferative disease. Allowable exceptions:

    1. Successfully treated cutaneous squamous cell or basal cell carcinoma
    2. Localized carcinoma in situ of the cervix
    3. Curatively treated malignancy (treatment terminated) > 5 years prior to screening
14. Subject has a history of listeriosis, histoplasmosis, untreated TB, persistent chronic infections, or recent active infections requiring hospitalization or treatment with intravenous (iv) anti-infectives within 30 days or oral anti-infectives within 14 days prior to the BL visit.
15. Subjects will be evaluated for latent TB infection with a PPD or QuantiFERON test and X-ray. Subjects with evidence for latent TB will not be enrolled but first assessed according to local guidelines.
16. Subject is known to have immune deficiency, history of Human Immunodeficiency Virus (HIV) or is otherwise severely immunocompromised.
17. Female subject who is pregnant or breast-feeding or considering becoming pregnant during the study or within 150 days after the last dose of study medication.
18. Men who are planning to father a child during the time they are included in the study
19. Subject has a history of clinically significant drug or alcohol usage in the last year.
20. Subject has a chronic widespread pain syndrome.
21. Subject is considered by the investigator, for any reason, to be an unsuitable candidate for the study.
22. Subject is unwilling to comply with the study protocol.
23. Screening clinical laboratory analyses show any of the following abnormal laboratory results:

    1. Aspartate transaminase (AST) or alanine transaminase (ALT) > 1.75 times upper limit of normal (ULN).
    2. Positive serum human chorionic gonadotropin (hCG).
    3. Positive tests for hepatitis B surface antigen (HBsAg) or hepatitis C serology indicative of current infection.
    4. Creatinine levels > 2x the ULN. If creatinine 1-2 times ULN, check GFR.
    5. Hemoglobin < 90 g/L.
    6. Absolute neutrophil count (ANC) < 1.5 x 10^3/microL.
    7. Serum total bilirubin > 1.5 mg/dL (>26 micromol/L).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 812 (Actual)
Dates: Start 2012-12-14 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients in remission at week 24 from baseline according to CDAI | 24 weeks from BL
  Treatment Part 1: The primary efficacy outcome is the proportion of patients in remission at week 24 from BL according to CDAI
The proportion of patients in remission at week 24 after dose-reduction according to CDAI | 24 weeks after dose-reduction
  Treatment Part 2: The primary efficacy outcome is the proportion of patients in remission according to CDAI, at the time point 24 weeks after the dose was first reduced
The radiographic progression of total Sharp van der Heijde score after 48 weeks from baseline | 48 weeks from BL
  The primary efficacy outcome is the progression of total Sharp van der Heijde score after 48 weeks from BL

CONTACTS AND LOCATIONS:
Overall Officials: Ronald van Vollenhoven, MD, Prof., Principal Investigator — The Karolinska Institute
Locations (30):
- Denmark (7):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
  - Silkeborg University Clinic, Silkeborg
  - Svendborg Hospital OUH, Svendborg
  - University Hospital of Southern Denmark, Sønderborg
- Finland (4):
  - Helsinki University Central Hospital, Helsinki
  - Central Finland Central Hospital, Jyväskylä
  - Kuopio University Hospital, Kuopio
  - Tampere University Hospital, Tampere
- Landspitali University Hospital, Reykjavik, Iceland
- Reade, Amsterdam, Netherlands
- Norway (5):
  - Ålesund Hospital, Ålesund
  - Haukeland University Hospital, Bergen
  - Diakonhjemmet Hospital, Oslo
  - University Hospital of North Norway, Tromsø
  - St. Olav's Hospital, Trondheim
- Sweden (12):
  - Falu Hospital, Falun
  - Sahlgrenska University Hospital, Gothenburg
  - The Karolinska University Hospital, Huddinge
  - Linköping University Hospital, Linköping
  - Skåne University Hospital, Lund
  - Skåne University Hospital, Malmo
  - Örebro University Hospital, Örebro
  - The Karolinska University Hospital, Solna
  - Academic Specialist Center, Stockholm
  - The Karolinska Institutet, Stockholm
  - Uppsala University Hospital, Uppsala
  - Västmanlands Hospital, Västerås

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lend K, Twisk JW, Kumar N, Dijkshoorn B, Lampa J, Rudin A, Hetland ML, Uhlig T, Nordstrom D, Ostergaard M, Gudbjornsson B, Sokka-Isler T, Grondal G, Horslev-Petersen K, Nurmohamed MT, Frostegard J, van Vollenhoven RF. Glucocorticoid treatment in early rheumatoid arthritis is independently associated with increased PCSK9 levels: data from a randomised controlled trial. RMD Open. 2025 Jun 5;11(2):e005129. doi: 10.1136/rmdopen-2024-005129. PMID 40480650
- [Derived] Lend K, Lampa J, Padyukov L, Hetland ML, Heiberg MS, Nordstrom DC, Nurmohamed MT, Rudin A, Ostergaard M, Haavardsholm EA, Horslev-Petersen K, Uhlig T, Sokka-Isler T, Gudbjornsson B, Grondal G, Frazzei G, Christiaans J, Wolbink G, Rispens T, Twisk JWR, van Vollenhoven RF. Association of rheumatoid factor, anti-citrullinated protein antibodies and shared epitope with clinical response to initial treatment in patients with early rheumatoid arthritis: data from a randomised controlled trial. Ann Rheum Dis. 2024 Nov 14;83(12):1657-1665. doi: 10.1136/ard-2024-226024. PMID 39079894
- [Derived] Dubovyk V, Vasileiadis GK, Fatima T, Zhang Y, Kapetanovic MC, Kastbom A, Rizk M, Soderbergh A, Zhao SS, van Vollenhoven RF, Hetland ML, Haavardsholm EA, Nordstrom D, Nurmohamed MT, Gudbjornsson B, Lampa J, Ostergaard M, Heiberg MS, Sokka-Isler T, Grondal G, Lend K, Horslev-Petersen K, Uhlig T, Rudin A, Maglio C. Obesity is a risk factor for poor response to treatment in early rheumatoid arthritis: a NORD-STAR study. RMD Open. 2024 Apr 4;10(2):e004227. doi: 10.1136/rmdopen-2024-004227. PMID 38580350
- [Derived] Ostergaard M, van Vollenhoven RF, Rudin A, Hetland ML, Heiberg MS, Nordstrom DC, Nurmohamed MT, Gudbjornsson B, Ornbjerg LM, Boyesen P, Lend K, Horslev-Petersen K, Uhlig T, Sokka T, Grondal G, Krabbe S, Lindqvist J, Gjertsson I, Glinatsi D, Kapetanovic MC, Aga AB, Faustini F, Parmanne P, Lorenzen T, Giovanni C, Back J, Hendricks O, Vedder D, Rannio T, Grenholm E, Ljosa MK, Brodin E, Lindegaard H, Soderbergh A, Rizk M, Kastbom A, Larsson P, Uhrenholt L, Just SA, Stevens DJ, Bay Laurbjerg T, Bakland G, Olsen IC, Haavardsholm EA, Lampa J; NORD-STAR study group. Certolizumab pegol, abatacept, tocilizumab or active conventional treatment in early rheumatoid arthritis: 48-week clinical and radiographic results of the investigator-initiated randomised controlled NORD-STAR trial. Ann Rheum Dis. 2023 Oct;82(10):1286-1295. doi: 10.1136/ard-2023-224116. Epub 2023 Jul 9. PMID 37423647
- [Derived] Stockfelt M, Lundell AC, Hetland ML, Ostergaard M, Uhlig T, Heiberg MS, Haavardsholm EA, Nurmohamed MT, Lampa J, Nordstrom D, Petersen KH, Gudbjornsson B, Grondal G, Aldridge J, Andersson K, Blennow K, Zetterberg H, van Vollenhoven R, Rudin A. Plasma interferon-alpha is associated with double-positivity for autoantibodies but is not a predictor of remission in early rheumatoid arthritis-a spin-off study of the NORD-STAR randomized clinical trial. Arthritis Res Ther. 2021 Jul 13;23(1):189. doi: 10.1186/s13075-021-02556-1. PMID 34256800
- [Derived] Hetland ML, Haavardsholm EA, Rudin A, Nordstrom D, Nurmohamed M, Gudbjornsson B, Lampa J, Horslev-Petersen K, Uhlig T, Grondal G, Ostergaard M, Heiberg MS, Twisk J, Lend K, Krabbe S, Hyldstrup LH, Lindqvist J, Hultgard Ekwall AK, Gron KL, Kapetanovic M, Faustini F, Tuompo R, Lorenzen T, Cagnotto G, Baecklund E, Hendricks O, Vedder D, Sokka-Isler T, Husmark T, Ljosa MA, Brodin E, Ellingsen T, Soderbergh A, Rizk M, Olsson AR, Larsson P, Uhrenholt L, Just SA, Stevens DJ, Laurberg TB, Bakland G, Olsen IC, van Vollenhoven R; NORD-STAR study group. Active conventional treatment and three different biological treatments in early rheumatoid arthritis: phase IV investigator initiated, randomised, observer blinded clinical trial. BMJ. 2020 Dec 2;371:m4328. doi: 10.1136/bmj.m4328. PMID 33268527
- [Derived] Glinatsi D, Heiberg MS, Rudin A, Nordstrom D, Haavardsholm EA, Gudbjornsson B, Ostergaard M, Uhlig T, Grondal G, Horslev-Petersen K, van Vollenhoven R, Hetland ML. Head-to-head comparison of aggressive conventional therapy and three biological treatments and comparison of two de-escalation strategies in patients who respond to treatment: study protocol for a multicenter, randomized, open-label, blinded-assessor, phase 4 study. Trials. 2017 Apr 4;18(1):161. doi: 10.1186/s13063-017-1891-x. PMID 28376912
- Available data/document: Study Protocol — http://www.biomedcentral.com/search?query=glinatsi&searchType=publisherSearch — Publication of the protocol. Glinatsi et al. Trials (2017) 18:161